CLINICAL TRIAL: NCT05468749
Title: A Phase 1 Study to Assess the Effect of Moderate Renal Impairment on the Pharmacokinetics of CTP-543 (Deuruxolitinib Phosphate)
Brief Title: Study to Assess the Effect of Renal Impairment on the Pharmacokinetics of CTP-543
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: CP543.1014
Record Dates: First submitted 2022-06-30; First posted 2022-07-21 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Renal Impairment
Keywords: CTP-543
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTP-543 Treatment (Experimental)
  Interventions: Drug: CTP-543

INTERVENTIONS:
Drug: CTP-543 — Single 12 mg oral dose administered on Day 1

SUMMARY:
This is an open-label, single-dose, sequentially designed, single-period study to determine the effect of moderate renal impairment on the pharmacokinetics (PK) of CTP-543 and its major metabolites following administration of a single 12 mg oral dose of CTP-543.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females aged 18-75
* Body mass index (BMI) ≥ 18.0 and ≤ 42.0 kg/m2 at the time of screening
* If of reproductive age, willing and able to use a medically highly effective form of birth control 30 days prior to first dose, during the study and for 30 days following last dose of study medication
* Capable of giving informed consent and complying with study procedures

Additional Inclusion Criteria for Subjects with Renal Impairment:

* eGFR of 30-59 mL/minute/1.73 m2 as calculated by the MDRD equation
* No clinically significant change in disease status within the last 30 days before screening
* The subject must have a condition consistent with renal impairment and associated symptoms, but otherwise be determined to be in good health in the opinion of the Investigator
* Concomitant medications to treat underlying disease states or medical conditions related to renal impairment are allowed with the exception of strong CYP3A4 inhibitors and inducers

Exclusion Criteria:

* History of any clinically significant medical condition, psychiatric disease, social condition, or illness that might confound the results of the study or poses an additional risk to the subject by their participation in the study
* Known history of any gastrointestinal surgery or any condition possibly affecting drug absorption
* History of prolonged QT syndrome or a QTc interval with Fridericia's correction (QTcF) > 470 msec for males or QTcF > 480 msec for females at Screening visit
* Positive for human immunodeficiency virus, Hepatitis B virus, or Hepatitis C virus
* Females who are nursing or pregnant prior to drug administration
* Positive results for coronavirus infection (COVID-19) at screening or check-in
* Positive drugs of abuse or alcohol results at screening or check in (Day -1)

Additional Exclusion Criteria for Subjects with Renal Impairment:

* History of renal transplant
* Significant bleeding diathesis that could preclude multiple venipuncture or deep intramuscular injections
* Acute or exacerbating renal disease
* History of drugs of abuse or alcohol misuse within 6 months prior to screening
* Poorly controlled Type 1 or Type 2 diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Single dose PK exposure: Maximum observed concentration (Cmax) | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48 hours post-dose
  Maximum concentration, obtained directly from the observed concentration versus time data.
Single dose PK exposure: Area Under the Concentration-Time Curve from time zero to the time of the last observed/measured non-zero concentration (AUC0-t) | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48 hours post-dose
  Area under the concentration-time curve from time zero (pre-dose) to time of last measurable concentration (calculated by linear-log trapezoidal summation)
Single dose PK exposure: Area Under the Concentration-Time Curve from time 0 extrapolated to infinity (AUC0-inf) | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48 hours post-dose
  Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinity, calculated by linear-log trapezoidal summation and extrapolated to infinity by addition of the last quantifiable concentration divided by the elimination rate constant

SECONDARY OUTCOMES:
Assessment of Safety and Tolerability following administration of CTP-543 | Screening (within 21 days prior to Day 1) through follow-up (7 to 10 days after final drug)
  Number of adverse events, including abnormal clinical laboratory findings, abnormal physical examinations, abnormal ECGs and abnormal vital signs tabulated for each subject

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee